CLINICAL TRIAL: NCT00641342
Title: Prevention of Parastomal Hernia by Primary Mesh Insertion: a Randomized Double-blinded Controlled Multi-centre Study.
Brief Title: Prevention of Parastomal Hernia by Primary Mesh Insertion
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Lack of recruitment from different study sites and due to structural changes in the included centers
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: Aarhus University Hospital (Other); Hvidovre University Hospital (Other); Copenhagen University Hospital at Herlev (Other); Esbjerg Hospital - University Hospital of Southern Denmark (Other); Hillerod Hospital, Denmark (Other); Vejle Hospital (Other); Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Ismail Gögenur, Dr, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PMPC
Record Dates: First submitted 2008-03-18; First posted 2008-03-24 (Estimated); Last update posted 2014-02-07 (Estimated); Status verified 2008-03

CONDITIONS: Parastomal Hernia
Keywords: Parastomal hernia; Onlay mesh; Sublay mesh; Pain; Health questionnaire
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- onlay mesh (Active Comparator)
  Interventions: Device: onlay mesh
- sublay mesh (Active Comparator)
  Interventions: Device: onlay mesh
- no mesh (No Intervention)

INTERVENTIONS:
Device: onlay mesh — StomaMesh (Precut heavyweight polypropylene mesh) Vypro Mesh (lightweight Prolene and vicryl mesh)
  Arms: onlay mesh; sublay mesh

SUMMARY:
Approximately 1/3 of patients with a permanent end-colostomy will experience a hernia around the stoma. In some cases these problems result in the need of surgical correction and the risk of recurrent hernia after operative intervention is regrettably high. Preliminary investigations suggest a role for primary mesh placement to prevent parastomal hernia. The use of a mesh as a preventive measure is a safe procedure. This study will focus on the effect of primary mesh placement (two different operative procedures are used) compared to patients without mesh placement.

ELIGIBILITY:
Inclusion Criteria:

* Permanent end-colostomy after surgery for rectosigmoid cancer with extirpation or Hartmann's procedure.

Exclusion Criteria:

* ASA > 3
* Acute surgery
* Known immune deficiency
* Surgery with insertion of foreign body (orthopaedic prosthesis, mechanical or bio-logical heart valve etc.) within the last 3 months.
* Pregnancy
* Known inflammatory bowel disease
* Lack of written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2007-03; Primary Completion 2015-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Parastomal hernia verified by CT-scan | one year after surgery, reassessed after 2, 3 and 5 years

SECONDARY OUTCOMES:
Clinically detected parastomal hernia | one year after surgery, reassessed after 2, 3 and 5 years
Pain | one year after surgery, reassessed after 2, 3 and 5 years
Disease specific and general health questionnaire | one year after surgery, reassessed after 2, 3 and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Ismail Gögenur, Principal Investigator — University Hospital of Copenhagen, GEntofte
Locations (2):
- Denmark (2):
  - Copenhagen University Hospital, Hvidovre, Hvidovre, Copebhagen
  - Copenhagen University Hospital, Gentofte, Hellerup, Copenhagen